CLINICAL TRIAL: NCT06905756
Title: Compartive Effect of Accelerated Rehabilitation and Eccentric Strengthing Exercises on Patient With Achilles Tendinopathy
Brief Title: Comparative Effect of Accelerated Rehabilitation and Eccentric Strengthening Exercises on Patients With AT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall23/788
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Achilles Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated rehabilitation (Experimental)
  Interventions: Diagnostic Test: Accelerated rehabilitation
- Eccentric strengthening exercises (Experimental)
  Interventions: Combination Product: Eccentric strengthening exercises

INTERVENTIONS:
Diagnostic Test: Accelerated rehabilitation — 15 subjects in group A will be receiving Accelerated Rehabilitation protocol alongwith baseline treatment. Accelerated rehabilitation consisting of three phases, following 12 week exercise regime. Pain reduction, mobility, strengthening, and functional recovery are part of the accelerated rehabilitation protocol for Achilles tendinopathy. Ice, TENS, range-of-motion exercises, isometric calf contractions, and a progressive transition to full weight-bearing based are the mainstays of Phase 1 (Weeks 1-4). Phase 2 (Weeks 5-8) focuses on balance training, resistance band exercises, and seated and standing calf raises as well as light functional workouts like cycling or walking. Phase 3 (Weeks 9-12) progresses to sport-specific and endurance exercises like swimming or running after including plyometric drills, eccentric heel drops, and advanced strengthening. Each exercise will be performed under supervision of skilled physiotherapist for 2 times daily, 2 sets of 5 repetitions.
  Arms: Accelerated rehabilitation
Combination Product: Eccentric strengthening exercises — Group B will be receiving eccentric strengthening exercises alongwith baseline treatment. Techniques of Curwin, Stanish et al will be used for eccentric training. For every exercise, participants do three sets of 15 repetitions, with a 30-second break in between. Weight is added gradually to enhance resistance (5-10 lbs or more, depending on tolerance). The eccentric strengthening regimen for Achilles tendinopathy advances every week. Participants use both feet without dorsiflexion to perform eccentric contractions in Week 1. By Week 3, the focus of the workouts is on the injured foot in maximum dorsiflexion. In Week 4, 10% body weight resistance is introduced, and in Week 5, an extra 5-10 pounds. From Week 6 to Week 8, resistance rises every two weeks. From Weeks 9 to 12, functional motions like hopping, single-leg heel drops, and sport-specific drills are incorporated, all of which are customized to meet individual goals.
  Arms: Eccentric strengthening exercises

SUMMARY:
A common overuse injury to the Achilles tendon, Achilles tendinopathy frequently causes pain, restricted range of motion, and functional impairment.

DETAILED DESCRIPTION:
The purpose of this randomized clinical research is to evaluate the benefits of eccentric strengthening exercises and rapid rehabilitation on Achilles tendinopathy patients. Using techniques including TENS, isometric exercises, balance training, and endurance exercises, the 12-week accelerated rehabilitation program emphasizes pain management, mobility restoration, and functional recovery through incremental phases. However, in order to improve tendon strength and resilience, eccentric strengthening entails progressively raising resistance and functional loading. Both approaches are backed by earlier research but lack direct comparison in terms of effectiveness. This study will open the door for more research and improve rehabilitation techniques worldwide by adding to the expanding corpus of material on Achilles tendinopathy care.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age greater than 18 years, clinically diagnosed with Achilles tendinopathy.
* Participants that are clinically diagnosed with Achilles tendinopathy.
* Duration of symptoms or pain for more than 1 month.
* Positive clinical tests, such as Thompson test, confirming Achilles tendinopathy.
* Tenderness to palpation along the Achilles tendon or localized pain during activity.
* Patients with a history of overuse injuries related to repetitive activities, such as running or jumping.

Exclusion Criteria:

* Following participants will be excluded from this study:
* Presence of systemic conditions such as rheumatoid arthritis, diabetes, or other inflammatory or neuromuscular disorders.
* History of complete Achilles tendon rupture or previous surgical intervention on the affected tendon.
* Patients with other lower limb injuries or conditions (e.g., fractures, ligament tears) that could interfere with Achilles tendinopathy treatment.
* Severe tendon degeneration or calcification confirmed by imaging, unsuitable for rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale | 12 Months
  The Pain Scale has a numerical rating system (NRS) with 11 points, with 0 denoting no pain and 10 denoting the most excruciating pain. The following categories apply to scores:
  0= denotes no pain 1-3= mild pain 4-6=moderate pain 7-10= severe pain.(12)
WHOQOL (world health organization and quality of life) | 12 Months
  The WHOQOL uses 26 questions to calculate quality of life across the four domains. Each item is scored on a 5-point Likert scale (1 to 5), where higher scores indicate a better quality of life, lower score indicate, poor quality of life. Average total score for healthy populations is about 90.
  0-20 = Poor Quality of Life 21-40 = Moderate Quality of Life 41-60 = Good Quality of Life 61-80 or greater than 80 = Very Good Quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Punjab Social Security Health Management Hospital Manga Raiwind, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No